CLINICAL TRIAL: NCT04313660
Title: Anlotinib In Combination With PD-1/L1 Inhibitor As Sequential Therapy of Thoracic Radiotherapy After Induction Chemotherapy For Extensive-Stage Small Cell Lung Cancer:A Single Arm Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVATAR
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: NSCLC; Anlotinib; PD-1/L1 Inhibitor
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib In Combination With PD-1/L1 Inhibitor (Experimental)
  Interventions: Drug: Anlotinib In Combination With PD-1/L1 Inhibitor

INTERVENTIONS:
Drug: Anlotinib In Combination With PD-1/L1 Inhibitor — At the end of chest radiotherapy (c2d1), the simultaneous administration of androtinib hydrochloride capsule and PD-1 / L1 inhibitor was started. L
  Arotinib hydrochloride capsule, 12 mg, Po, QD, was taken orally for two weeks, one week, three weeks as a cycle, completed in the first 14 days until the disease progress;
  Durvalumab injection, 1500mg, IV, once every three weeks, completed on the first day until the disease progresses.
  Tetraprizumab injection, 240mg, IV, once every three weeks, completed on the first day until the disease progresses.
  The choice of durvalumab / trepril mAb was at the discretion of the researchers.

SUMMARY:
Anlotinib In Combination With PD-1/L1 Inhibitor As Sequential Therapy of Thoracic Radiotherapy After Induction Chemotherapy For Extensive-Stage Small Cell Lung Cancer:A Single Arm Study

ELIGIBILITY:
Inclusion Criteria:

1. The subjects volunteered to join the study and signed the informed consent form. They had good compliance and cooperated with the follow-up;
2. Patients between 18-75 years old;
3. Extensive small cell lung cancer confirmed by histopathology (according to Veterans Administration lung study group, Valg stage) and did not progress after 4-6 cycles (21 days as a cycle) of first-line standard chemotherapy platinum combined with etoposide [complete remission (CR), partial remission (PR) or stable (SD) according to recist1.1 standard];
4. The time interval between the first TRT and the end of the last chemotherapy should be less than or equal to 6 weeks;
5. The life expectancy shall be at least 3 months;
6. ECoG score: 0-1

Exclusion Criteria:

1. Small cell lung cancer patients with other pathological types of tumor species;
2. Patients with pathological fracture in bone metastasis of small cell lung cancer;
3. Patients with central nervous system metastasis;
4. Patients who have received chest radiotherapy before;
5. Patients who have used vasotargeted drugs (such as bevacizumab, sunitinib, etc.) including enrotinib and immunosuppressive agents before;
6. Imaging (CT or MRI) showed that the distance between the tumor focus and the large blood vessel was less than or equal to 5 mm, or there was a central tumor invading the local large blood vessel, or there was an obvious cavitary or necrotic tumor in the lung;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
progress free survival(PFS) | 1 year
  the period from the beginning of treatment to the observation of disease progress or death for any reason

SECONDARY OUTCOMES:
Overall survival(OS) | 1 year
  Time from randomization to death for any reason. The last follow-up time is usually calculated as the time of death for the subjects who have lost the visit before death